CLINICAL TRIAL: NCT01544309
Title: Study on Effect of Highly Potent Statins on Lipid Lowering Effect and Glucose Metabolism in Hypercholesterolemia Patients With Diabetes Mellitus
Brief Title: LIpid Lowering With Highly Potent Statins in Hyperlipidaemia With Type 2 Diabetes patiENts
Acronym: LISTEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Listen Trial Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0059
Record Dates: First submitted 2012-02-23; First posted 2012-03-05 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Hypercholesterolemia With Concomitant Type 2 Diabetes
MeSH Terms: interventions — Atorvastatin; Rosuvastatin Calcium

ARMS (2):
- Atorvastatin administration group (Experimental)
  Interventions: Drug: Atorvastatin
- Rosuvastatin administration group (Experimental)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 10 mg (atorvastatin 10 mg tablet x 1 or atorvastatin 5 mg tablet x 2), orally,once daily for 12 months.
  (When not reach the LDL-C level of target in the Japan Atherosclerosis Society [JAS] Guidelines [GL] after 3 months, had the atorvastatin [ATV] dose of 20 mg.)
  Other Names: Lipitor
  Arms: Atorvastatin administration group
Drug: Rosuvastatin — Rosuvastatin 5 mg (rosuvastatin 5 mg tablet x1 or rosuvastatin 2.5 mg tablet x 2), orally, once daily for 12 months.
  (When not reach the LDL-C level of target in JAS GL after 3 months, had the rosuvastatin [RSV] dose of 10 mg.)
  Other Names: Crestor
  Arms: Rosuvastatin administration group

SUMMARY:
The purpose of this study is to compare the effect of rosuvastatin and atorvastatin on lipid lowering effect and glucose metabolism in hypercholesterolemia patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Hypercholesterolemia patients

   • Patients who have not achieved the target control levels of LDL-C in the "Japan Atherosclerosis Society Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2007"
2. Type 2 diabetes patients

   * Patients diagnosed with type 2 diabetes and receiving diet therapy, exercise therapy, or medication
   * Patients who received constant therapy for three months before registration and have no plan for therapy change
   * Patients with kept HbA1c level (Japan Diabetes Society [JDS] level) of less than 7.0% (or, National Glycohemoglobin Standardization Program [NGSP] level of less than 7.4%) within three months before registration
   * Patients receiving or not receiving medication at present
3. Patients giving voluntary written consent to participate in the study
4. Male or female patients at 20 years or older

Exclusion Criteria:

1. Patients who administered rosuvastatin, atorvastatin or ezetimibe within three month at the registration
2. Patients with severe hypertension (systolic blood pressure [SBP] ≥ 180 mmHg or diastolic blood pressure [DBP] ≥ 110 mmHg)
3. Patients with type 1 diabetes
4. Patients judged to have familial hypercholesterolemia
5. Patients with a serum triglyceride level of ≥ 400 mg/dL
6. Patients who had the onset of cardiovascular or cerebrovascular disease within three months
7. Patients with serious heart failure (NYHA classification III - IV)
8. Patients with a history of hypersensitivity to statins
9. Patients with a history of drug-induced myopathy
10. Patients with severe complication of diabetes
11. Patients receiving insulin
12. Patients with serious liver or kidney disease
13. Patients with serious concurrent disease such as malignancy, or patients with severely limited lifespan
14. Patients who are or may be pregnant
15. Patients judged by the investigators to be ineligible for participation in the study for any other reason

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1049 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, Ph.D, Study Chair — Department of Cardiovascular Medicine, Faculty of Life Sciences, Kumamoto University
Locations (133):
- Japan (133):
  - Hiramitsu Heart Clinic, Nagoya, Aichi Pref.
  - Honjo Daiichi Hospital, Yurihonjō, Akita Pref.
  - Iryouhoujin Syadan Yanagisawakai Yanagisawa Iin, Matsudo, Chiba Pref.
  - Matsuno Medical Clinic, Iyo Gun, Ehime Pref.
  - Ishite Matsumoto Naika Junkanki Clinic, Matsuyama, Ehime Pref.
  - Ehime Medical CO OP Izumigawa Clinic, Niihama, Ehime Pref.
  - Fukui Chuoh Clinic, Fukui, Fukui Pref.
  - Fukuoka City Medical Association Hospital, Fukuoka, Fukuoka Pref.
  - Matsumoto Clinic, Fukuoka, Fukuoka Pref.
  - Saku Hospital, Fukuoka, Fukuoka Pref.
  - Soejima Medical Clinic, Fukuoka, Fukuoka Pref.
  - Takei's Clinic Internal Medicine, Fukuoka, Fukuoka Pref.
  - Nakamura Cardiovascular Clinic, Itoshima, Fukuoka Pref.
  - Morizono Naika, Kitakyushu, Fukuoka Pref.
  - Seino Internal Medicine Clinic, Kōriyama, Fukushima Pref.
  - Yasue Naika, Gifu, Gifu City
  - Kawade Iin, Gifu, Gifu Pref.
  - Hashimoto Naika Clinic, Gifu, Gifu Pref.
  - Iinuma Iin, Gifu, Gifu Pref.
  - Ishimura Clinic, Gifu, Gifu Pref.
  - Kawai Clinic, Gifu, Gifu Pref.
  - Niimi Clinic, Gifu, Gifu Pref.
  - Takai Clinic, Gifu, Gifu Pref.
  - Kobayashi Internal Medicine, Kakamigahara, Gifu Pref.
  - Horibe Clinic, Motosu, Gifu Pref.
  - Kondo Cardiovascular Clinic, Ōgaki, Gifu Pref.
  - Yoshida Naika, Ōgaki, Gifu Pref.
  - Kogure Clinic, Maebashi, Gunma Pref.
  - Nakano Clinic, Shibukawa, Gunma Pref.
  - Yoshii Central Clinic, Takasaki, Gunma Pref.
  - Shigenobu Clinic, Miyoshi, Hiroshima Pref.
  - Takahashi Kiyohito Clinic, Hakodate, Hokkaido Pref.
  - Hokuto Internal Medicine Clinic, Sapporo, Hokkaido Pref.
  - Katsuya Clinic, Amagasaki, Hyogo Pref.
  - Nakatani Hospital, Himeji, Hyogo Pref.
  - Kosumo Clinic, Kako Gun, Hyogo Pref.
  - Harima Clinic, Kakogawa, Hyogo Pref.
  - Kusunose Clinic, Kobe, Hyogo Pref.
  - Yanagi Medical Clinic, Hakusan, Ishikawa Pref.
  - Okyozuka Clinic, Ishikawa Gun, Ishikawa Pref.
  - Doniwa Clinic, Kanazawa, Ishikawa Pref.
  - Wakasa Medical Clinic, Kanazawa, Ishikawa Pref.
  - Association Medical Corporation Neurology Internal Medicine Kanamori Clinic, Iwate Gun, Iwate Pref.
  - Medical Corporation Kuon-kai Kamata Medical Clinic, Morioka, Iwate Pref.
  - Kagawa Clinic, Marugame, Kagawa Pref.
  - Hasegawa Outpatients Clinic for Cardiovascular Disease, Takamatsu, Kagawa Pref.
  - Tempozan Naika Clinic, Kagoshima, Kagoshima Pref.
  - Kashiwagi Clinic, Ayase, Kanagawa Pref.
  - Hayashi Diabetes Clinic, Chigasaki, Kanagawa Pref.
  - Takada Internal Medicine Clinic, Hiratsuka, Kanagawa Pref.
  - Iroden Clinic, Kamakura, Kanagawa Pref.
  - Nagasu Clinic, Kamakura, Kanagawa Pref.
  - Kobayashi Hospital, Odawara, Kanagawa Pref.
  - Hakuai Iin, Sagamihara, Kanagawa Pref.
  - Yamamoto Clinic, Sagamihara, Kanagawa Pref.
  - Arima Clinic, Yokohama, Kanagawa Pref.
  - Kikuchi Clinic, Yokohama, Kanagawa Pref.
  - Miho cho Cardiovascular Medical Clinic, Yokohama, Kanagawa Pref.
  - Minamisawa Clinic, Yokohama, Kanagawa Pref.
  - Shimokurata Heart Clinic, Yokohama, Kanagawa Pref.
  - Yokohama Sotetsu Bldg. Clinic of Internal Medicine, Yokohama, Kanagawa Pref.
  - Jinnouchi Clinic Diabetes Care Center, Kumamoto, Kumamoto Pref.
  - Maki Cardiovascular Clinic, Kumamoto, Kumamoto Pref.
  - Munakata Clinic, Kumamoto, Kumamoto Pref.
  - Terao Hospital, Kumamoto, Kumamoto Pref.
  - Higashi Diabetes and Cardiovascular Clinic, Tamana, Kumamoto Pref.
  - Matsuo Clinic, Tamana, Kumamoto Pref.
  - Miyagi Clinic Cardiovascular Medicine, Yatsushiro, Kumamoto Pref.
  - Asamoto Internal Medical Clinic, Kyoto, Kyoto Pref.
  - Ijinkai Takeda General Hospital, Kyoto, Kyoto Pref.
  - Koseikai Clinic, Kyoto, Kyoto Pref.
  - Sakabe International Clinic, Kyoto, Kyoto Pref.
  - Takenaka Clinic, Kyoto, Kyoto Pref.
  - Tegoshi Clinic, Kyoto, Kyoto Pref.
  - Sawai Naika Iin, Kyōtanabe, Kyoto Pref.
  - Iwasaki Hospital, Tsu, Mie Pref.
  - Ishikawa Clinic, Miyazaki, Miyazaki Pref.
  - Yokota Naika, Miyazaki, Miyazaki Pref.
  - Etou Clinic, Nichinan, Miyazaki Pref.
  - Kawano Clinic, Nichinan, Miyazaki Pref.
  - Yamaguchi Clinic, Nichinan, Miyazaki Pref.
  - Hasegawa Clinic, Nakano City, Nagano Pref.
  - Nara Prefectural Gojo Hospital, Gojō, Nara Pref.
  - Fujii Internal Medicine Clinic, Kashihara, Nara Pref.
  - Matsuoka Clinic, Kita Katsuragi Gun, Nara Pref.
  - Ote Clinic of Internal, Sakurai, Nara Pref.
  - Uchiyama Clinic, Jōetsu, Niigata Pref.
  - Inoue Clinic, Niigata, Niigata Pref.
  - Maeda Medical Clinic, Niigata, Niigata Pref.
  - Nishimura Clinic, Fujiidera, Osaka Pref.
  - Shoseikai Matsuda Iin, Fujiidera, Osaka Pref.
  - Ikeda Clinic, Higashiosaka, Osaka Pref.
  - Kanazawa Clinic, Izumi, Osaka Pref.
  - Fukuda Clinic, Osaka, Osaka Pref.
  - Jikuhara Clinic, Osaka, Osaka Pref.
  - Kawagishi-naika Clinic, Osaka, Osaka Pref.
  - Kinugawa Cardiology Clinic, Osaka, Osaka Pref.
  - Kubota Clinic, Osaka, Osaka Pref.
  - Masaki Clinic, Osaka, Osaka Pref.
  - Nanko Clinic, Osaka, Osaka Pref.
  - Osaka Ekisaikai Hospital, Osaka, Osaka Pref.
  - Tamatani Clinic, Osaka, Osaka Pref.
  - Hayashi Clinic, Sakai, Osaka Pref.
  - Nakao Medical Clinic, Sakai, Osaka Pref.
  - Saga Memorial Clinic, Saga, Saga Pref.
  - Enomoto Clinic, Ageo, Saitama Pref.
  - Asano Internal Medicine Clinic, Kawagoe, Saitama Pref.
  - Iryohojin Hogi Sinryojyo, Kawaguchi, Saitama Pref.
  - Tokutake Iin, Kawaguchi, Saitama Pref.
  - Medical Corporation Shibuya Clinic, Kumagaya, Saitama Pref.
  - Tanaka Medical Clinic, Saitama, Saitama Pref.
  - Yoshimura Eye&Internal Medical Clinic, Mishima, Shizuoka Pref.
  - Shizuoka Municipal Hospital, Shizuoka, Shizuoka Pref.
  - Takada Clinic, Tochigi, Tochigi Pref.
  - Murakami Clinic, Anan, Tokushima Pref.
  - Ota Clinic, Awa, Tokushima Pref.
  - Arizumi Clinic, Itano Gun, Tokushima Pref.
  - Yuki National Health Insurance Hospital of Minami Town, Kaifu Gun, Tokushima Pref.
  - Sekishinkan Hospital, Komatsushima, Tokushima Pref.
  - Iryohojin Tokujikai Tanaka Iin, Myozai Gun, Tokushima Pref.
  - Kensei Uchimachi Clinic, Tokushima, Tokushima Pref.
  - Yata Clinic, Yoshinogawa, Tokushima Pref.
  - Tokyo Center Clinic, Chuo Ku, Tokyo
  - Okudo Poly Clinic, Katsushika-ku, Tokyo
  - Nakano Sunbright Clinic, Nakano Ku, Tokyo
  - Sugawara Clinic, Nerima Ku, Tokyo
  - Tsurumachi Clinic, Setagaya Ku, Tokyo
  - Oda Clinic, Shinjuku Ku, Tokyo
  - Ishii Clinic, Tachikawa, Tokyo
  - Ayame Medical Clinic, Shimonoseki, Yamaguchi Pref.
  - Matsuda Medical Clinic, Shimonoseki, Yamaguchi Pref.
  - Mizumachi Medical Clinic, Shimonoseki, Yamaguchi Pref.
  - Kuroda Iin, Ōtsuki, Yamanashi Pref.

REFERENCES:
- [Derived] Ogawa H, Matsui K, Saito Y, Sugiyama S, Jinnouchi H, Sugawara M, Masuda I, Mori H, Waki M, Yoshiyama M, Watada H. Differences between rosuvastatin and atorvastatin in lipid-lowering action and effect on glucose metabolism in Japanese hypercholesterolemic patients with concurrent diabetes. Lipid-lowering with highly potent statins in hyperlipidemia with type 2 diabetes patients (LISTEN) study -. Circ J. 2014;78(10):2512-5. doi: 10.1253/circj.cj-14-0810. Epub 2014 Sep 2. PMID 25186922

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin Administration Group: Atorvastatin: Atorvastatin 10 mg (atorvastatin 10 mg tablet x 1 or atorvastatin 5 mg tablet x 2), orally,once daily for 12 months.
  (When not reach the LDL-C level of target in the Japan Atherosclerosis Society (JAS) Guidelines (GL) after 3 months, had the atorvastatin [ATV] dose of 20 mg.)
Period: Overall Study
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Started | 524 | 525
Completed | 504 | 514
Not Completed | 20 | 11
Not completed — Withdrawal by Subject | 12 | 7
Not completed — Protocol Violation | 2 | 1
Not completed — Physician Decision | 4 | 1
Not completed — Not performed pre-dose examination | 1 | 2
Not completed — Administered prohibit prior medication | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) - All participants who received at least 1 dose of open-label study drug except the ones who had no HbA1c or non-HDL-C data or a protocol deviation of the administration of study drugs.
Groups:
- Atorvastatin Administration Group: Atorvastatin: Atorvastatin 10 mg (atorvastatin 10 mg tablet x 1 or atorvastatin 5 mg tablet x 2), orally,once daily for 12 months.
  (When not reach the LDL-C level of target in JAS GL after 3 months, had the ATV dose of 20 mg.)
- Rosuvastatin Administration Group: Rosuvastatin: Rosuvastatin 5 mg (rosuvastatin 5 mg tablet x1 or rosuvastatin 2.5 mg tablet x 2), orally, once daily for 12 months.
  (When not reach the LDL-C level of target in JAS GL after 3 months, had the RSV dose of 10 mg.)
- Total: Total of all reporting groups
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group | Total
Number analyzed (Participants) | 504 | 514 | 1018
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.6) | 66.3 (11.6) | 66.4 (11.1)
Sex/Gender, Customized [Number; unit: participants]
  Male | 504 | 514 | 1018
Statin administration before entry [Number; unit: participants]
  Administered | 120 | 121 | 241
  Not administered | 384 | 393 | 777
Cardiovascular and Cerebrovascular events before entry [Number; unit: participants]
  With events | 103 | 103 | 206
  Without events | 401 | 411 | 812
Myocardial infarction [Number; unit: participants]
  With events | 7 | 7 | 14
  Without events | 497 | 507 | 1004
Angina pectoris [Number; unit: participants]
  With events | 31 | 31 | 62
  Without events | 473 | 483 | 956
Heart failure [Number; unit: participants]
  With events | 10 | 8 | 18
  Without events | 494 | 506 | 1000
Revascularization [Number; unit: participants]
  With events | 3 | 9 | 12
  Without events | 501 | 505 | 1006
Cardiac arrhythmias [Number; unit: participants]
  With events | 31 | 26 | 57
  Without events | 473 | 488 | 961
Cerebral haemorrhage [Number; unit: participants]
  With events | 3 | 6 | 9
  Without events | 501 | 508 | 1009
Cerebral infarction [Number; unit: participants]
  With events | 21 | 30 | 51
  Without events | 483 | 484 | 967
Transient ischaemic attack [Number; unit: participants]
  With events | 5 | 4 | 9
  Without events | 499 | 510 | 1009
Complications related to diabetes [Number; unit: participants]
  With diabetic complications | 49 | 67 | 116
  Without diabetic complications | 455 | 447 | 902
Diabetic retinopathy [Number; unit: participants]
  With diabetic retinopathy | 4 | 9 | 13
  Without diabetic retinopathy | 500 | 505 | 1005
Diabetic nephropathy [Number; unit: participants]
  With diabetic nephropathy | 13 | 21 | 34
  Without diabetic nephropathy | 491 | 493 | 984
Diabetic neuropathy [Number; unit: participants]
  With diabetic neuropathy | 23 | 23 | 46
  Without diabetic neuropathy | 481 | 491 | 972
Diabetic foot [Number; unit: participants]
  With diabetic foot | 0 | 1 | 1
  Without diabetic foot | 504 | 513 | 1017
Hypertension [Number; unit: participants]
  With hypertension | 307 | 338 | 645
  Without hypertension | 197 | 176 | 373
Non-high-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 169.0 (30.6) | 168.9 (35.8) | 168.9 (33.3)
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 139.6 (27.9) | 139.2 (31.9) | 139.4 (30.0)
HDL-C [Mean (Standard Deviation); unit: mg/dL] | 55.8 (14.6) | 54.1 (13.6) | 54.9 (14.1)
Total cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] | 224.8 (31.8) | 223.0 (36.0) | 223.9 (34.0)
Triglyceride (TG) [Mean (Standard Deviation); unit: mg/dL] | 149.6 (89.1) | 154.5 (137.1) | 152.1 (115.8)
Non-HDL-C/HDL-C ratio [Mean (Standard Deviation); unit: ratio] | 3.25 (1.07) | 3.36 (1.31) | 3.30 (1.20)
LDL-C/HDL-C ratio [Mean (Standard Deviation); unit: ratio] | 2.66 (0.81) | 2.73 (0.91) | 2.69 (0.86)
Free fatty acids (FFA) [Mean (Standard Deviation); unit: mEq/L] | 0.585 (0.297) | 0.584 (0.299) | 0.584 (0.298)
HbA1c [Mean (Standard Deviation); unit: % (NGSP value)] | 6.38 (0.59) | 6.40 (0.66) | 6.39 (0.63)
Blood glucose [Mean (Standard Deviation); unit: mg/dL] | 118.8 (27.0) | 119.1 (31.2) | 118.9 (29.2)
Insulin [Mean (Standard Deviation); unit: μU/mL] | 10.95 (18.66) | 12.57 (20.07) | 11.77 (19.39)
1,5-anhydro-D-glucitol (1,5-AG) [Mean (Standard Deviation); unit: μg/mL] | 15.40 (7.91) | 15.39 (8.10) | 15.40 (8.01)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Non-high-density Lipoprotein Cholesterol (HDL-C) Level
Time Frame: Baseline, and 12 months after administration
Population: Participants in full analysis set (FAS) except the ones who had no HDL-C data at 12 months.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 472 | 468
Percent change | -31.3 (19.1) | -32.8 (18.1)

2. Primary Outcome: Change in HbA1c Level
Time Frame: Baseline, 12 months after administration
Population: Participants in FAS except the ones who had no HbA1c data at 12 months.
Measure: Mean (Standard Deviation); unit: Amount of change (%)
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 472 | 468
Amount of change (%) | 0.120 (0.65) | 0.10 (0.67)

3. Secondary Outcome: Occurrence of Deterioration of Diabetic Treatment Status
Description: "Deterioration of diabetic treatment status" is defined as addition of new drug, increase in dosage, drug changes (therapy intensification), and deterioration in HbA1c of > 0.5%.
Time Frame: Baseline, 12 months after administration
Population: Full analysis set - All participants who received at least 1 dose of open-label study drug except the ones who had no HbA1c or non-HDL-C data or a protocol deviation of the administration of study drugs.
Measure: Number; unit: Participants
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 504 | 514
Participants
  Therapy intensification | 64 | 45
  Deterioration in HbA1c of > 0.5% | 177 | 162

4. Secondary Outcome: Number of Participants Stratified by Time to the Occurrence of Deterioration of Diabetic Treatment Status
Description: as for outcome 3
Time Frame: Baseline, 3, 6, 12 months after administration
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 504 | 514
participants
  Therapy intensification: 0-3 months | 20 | 14
  Therapy intensification: 3-6 months | 12 | 8
  Therapy intensification: 6-12 months | 32 | 23
  Other: 0-3 months | 6 | 5
  Other: 3-6 months | 5 | 5
  Other: 6-12 months | 8 | 6
  No deterioration | 421 | 453

5. Secondary Outcome: Percent Change in 1,5-AG Level
Description: An inverse relationship exists between mean change in 1,5-AG level and the mean rate of change when the degree of standard deviation is large, wherein the mean change is negative although the mean rate of change is positive or vice versa
Time Frame: Baseline, 3, 6, 12 months after administration and the end of study treatment（or at the occurrence of deterioration of diabetic treatment status）
Population: Participants in FAS except the ones who had no 1,5-AG data at 12 months.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 503 | 514
Percent change
  At 3 months | -1.6 (30.8) | 5.5 (72.6)
  At 6 months | -6.5 (35.8) | 2.6 (83.7)
  At 12 months | -3.8 (35.1) | 3.5 (98.0)

6. Secondary Outcome: Change in HbA1c Level
Time Frame: Baseline, 3, 6 months after administration and the end of study treatment （or at the occurrence of deterioration of diabetic treatment status）
Population: Full analysis set - All participants who received at least 1 dose of open-label study drug.
Measure: Mean (Standard Deviation); unit: Amount of change (%)
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 504 | 514
Amount of change (%)
  At 3 months | 0.05 (0.42) | 0.00 (0.50)
  At 6 months | 0.13 (0.57) | 0.12 (0.65)

7. Secondary Outcome: Percent Change in Blood Glucose Level (Fasting)
Time Frame: as for outcome 5
Population: Participants in FAS except the ones who had no blood glucose level data at 12 months.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 503 | 514
Percent change
  At 3 months | 3.3 (19.3) | 2.7 (25.0)
  At 6 months | 7.0 (24.1) | 5.9 (25.7)
  At 12 months | 4.6 (24.3) | 3.7 (26.1)

8. Secondary Outcome: Change in Blood Glucose Level (Fasting)
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Atorvastatin Administration Group: Atorvastatin 10 mg (atorvastatin 10 mg tablet x 1 or atorvastatin 5 mg tablet x 2), orally,once daily for 12 months.
  (When not reach the LDL-C level of target in JAS GL after 3 months, had the ATV dose of 20 mg.)
- Rosuvastatin Administration Group: Rosuvastatin 5 mg (rosuvastatin 5 mg tablet x1 or rosuvastatin 2.5 mg tablet x 2), orally, once daily for 12 months.
  (When not reach the LDL-C level of target in JAS GL after 3 months, had the RSV dose of 10 mg.)
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 503 | 514
mg/dL
  At 3 months | 2.6 (24.5) | 0.1 (31.2)
  At 6 months | 6.8 (30.2) | 4.3 (31.5)
  At 12 months | 3.6 (30.7) | 1.5 (35.0)

9. Secondary Outcome: Percent Change in Insulin Level
Description: An inverse relationship exists between mean change in insulin level and the mean rate of change when the degree of standard deviation is large, wherein the mean change is negative although the mean rate of change is positive or vice versa.
Time Frame: Baseline, 3, 6, 12 months after administration and the end of study treatment （or at the occurrence of deterioration of diabetic treatment status）
Population: Full analysis set - All participants who received at least 1 dose of open-label study drug
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 503 | 514
Percent change
  At 3 months | 40.7 (211.2) | 31.3 (166.4)
  At 6 months | 45.1 (193.9) | 35.5 (142.8)
  At 12 months | 17.4 (132.9) | 13.8 (148.1)

10. Secondary Outcome: Change From Baseline in Insulin Level
Description: as for outcome 9
Time Frame: as for outcome 9
Population: Full analysis set - All participants who received at least 1 dose of open-label study drug.
Measure: Mean (Standard Deviation); unit: μU/mL
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 503 | 514
μU/mL
  At 3 months | -0.10 (20.26) | -0.54 (18.56)
  At 6 months | 0.66 (18.63) | -0.44 (19.86)
  At 12 months | -1.50 (18.69) | -2.91 (19.02)
  Baseline Insulin level | 10.95 (18.66) | 12.57 (20.07)

11. Secondary Outcome: Frequency of Cardiovascular Events (Coronary Artery Disease, Heart Failure, Cerebrovascular Disease, Peripheral Artery Disease and Aortic Disease)
Time Frame: From the start of the treatment to the end of study treatment
Measure: Number; unit: Number of patients with any events
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 504 | 514
Number of patients with any events | 5 | 9

12. Secondary Outcome: Frequency of Serious Adverse Events (SAE)
Time Frame: Up to 12 months
Measure: Number; unit: Number of patients with SAE
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 506 | 516
Number of patients with SAE | 14 | 19

13. Secondary Outcome: Percent Changes in Lipids (LDL-C, HDL-C, TC, TG, Non-HDL-C/HDL-C Ratio, and FFA)
Time Frame: Baseline, 3, 6, 12 months after administration, the end of starting dose and the end of study treatment
Population: Participants in FAS except the ones who had no lipids level data at 12 months.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 504 | 514
Percent change
  LDL-C: at 3 months | -36.6 (19.2) | -39.2 (21.3)
  LDL-C: at 6 months | -35.6 (19.4) | -36.4 (21.8)
  LDL-C: at 12 months | -33.2 (21.5) | -34.7 (21.0)
  HDL-C: at 3 months | 4.1 (14.3) | 5.6 (13.9)
  HDL-C: at 6 months | 7.1 (15.1) | 8.2 (15.2)
  HDL-C: at 12 months | 4.9 (14.7) | 7.7 (15.9)
  TC: at 3 months | -24.7 (13.3) | -25.9 (14.3)
  TC: at 6 months | -23.5 (13.0) | -23.8 (14.9)
  TC: at 12 months | -22.7 (14.3) | -23.5 (14.0)
  TG at 3 months | -12.7 (38.0) | -11.0 (42.2)
  TG: at 6 months | -12.4 (45.9) | -11.9 (38.0)
  TG: at 12 months | -12.6 (62.2) | -15.9 (35.4)
  Non-HDL-C/HDL-C ratio: at 3 months | -34.8 (22.6) | -37.7 (20.2)
  Non-HDL-C/HDL-C ratio: at 6 months | -36.1 (19.4) | -37.2 (20.8)
  Non-HDL-C/HDL-C ratio: at 12 months | -33.1 (22.7) | -36.0 (20.7)
  FFA: at 3 months | 19.9 (87.8) | 25.9 (111.3)
  FFA: at 6 months | 13.8 (80.5) | 15.9 (88.9)
  FFA: at 12 months | 37.2 (125.3) | 34.8 (111.0)

14. Secondary Outcome: Percent Change in Non-HDL-C Level
Time Frame: Baseline, 3 and 6 months after administration, the end of starting dose and the end of study treatment
Population: Participants in FAS except the ones who had no non-HDL-C level data at 12 months.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 504 | 514
Percent change
  At 3 months | -33.8 (17.6) | -35.5 (18.4)
  At 6 months | -33.2 (16.6) | -33.5 (18.8)

15. Secondary Outcome: Percent Changes in Lipids and Inflammatory Marker (Hs-CRP) and Their Correlation
Description: Correlation between percent changes in lipids (LDL-C, HDL-C, non-HDL-C, TG, non-HDL-C/HDL-C ratio, LDL-C/HDL-C ratio, TC and FFA) and inflammatory marker (hs-CRP)
Time Frame: Baseline, 3, 6, 12 months after administration, the end of starting dose and the end of study treatment
Reporting Status: Not Posted

16. Secondary Outcome: Rate of Patients Who Have Reached the Target LDL-C Level Specified in Japan Atherosclerosis Society Guidelines (JASGL) 2007
Description: Percentage of participants achieving the target LDL-C levels <100 mg/dL for participants with history of coronary artery diseases (CAD) and <120 mg/dL for participants without history of CAD are presented.
Time Frame: 3 months after administration, the end of starting dose and the end of study treatment
Population: Full analysis set except participants who have reached the target LDL-C level specified at the treatment start
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 383 | 366
Percentage of participants
  At 3 months | 89.0 [85.5 to 92.0] | 89.9 [86.3 to 92.8]
  At the end of study treatment | 86.3 [82.5 to 89.6] | 87.5 [83.7 to 90.7]

17. Secondary Outcome: Change From Baseline in 1,5-AG Level
Description: as for outcome 5
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Number analyzed (Participants) | 503 | 514
μg/mL
  At 3 months | -0.51 (3.48) | -0.21 (3.77)
  At 6 months | -1.28 (4.23) | -0.94 (4.64)
  At 12 months | -0.88 (4.33) | -1.09 (4.66)
  Baseline 1,5-AG level | 15.40 (7.91) | 15.39 (8.10)

ADVERSE EVENTS:
Time Frame: At the start of the treatment, 3, 6, and 12 months after administration
Description: Analyzed: Safety analysis set - all participants who received at least 1 dose of open-label study drug.
Arm/Group | Atorvastatin Administration Group | Rosuvastatin Administration Group
Serious Adverse Events (participants affected / at risk) | 14/506 | 19/516
Other Adverse Events (participants affected / at risk) | 87/506 | 88/516
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin Administration Group (N=506) | Rosuvastatin Administration Group (N=516)
Pneumonia (Infections and infestations) | 1 (1) | 2
Diverticulitis (Infections and infestations) | 0 | 1
Nocardiosis (Infections and infestations) | 1 | 0
Keratitis fungal (Infections and infestations) | 1 | 0
Large intestine carcinoma (Musculoskeletal and connective tissue disorders) | 1 | 1
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Thrombosis in device (General disorders) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin Administration Group (N=506) | Rosuvastatin Administration Group (N=516)
Nasopharyngitis (Infections and infestations) | 13 | 15
Bronchitis (Infections and infestations) | 3 | 3
Cystitis (Infections and infestations) | 1 | 5
Pneumonia (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 2 | 2
Pharyngitis (Infections and infestations) | 1 | 2
Rhinitis (Infections and infestations) | 0 | 2
Oral herpes (Infections and infestations) | 1 | 1
Body tinea (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 1
Pertussis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Purulence (Infections and infestations) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 3
Goitre (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 1 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Illusion (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Dizziness (Nervous system disorders) | 5 | 6
Hypoaesthesia (Nervous system disorders) | 2 | 2
Dizziness postural (Nervous system disorders) | 1 | 2
Cerebral infarction (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness exertional (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Blepharitis (Eye disorders) | 0 | 1
Blepharospasm (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Corneal erosion (Eye disorders) | 1 | 0
Posterior capsule opacification (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 1
Palpitations (Cardiac disorders) | 3 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Essential hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 14
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 3 | 1
Gastritis (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 2
Cholangitis (Hepatobiliary disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 4 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Atonic urinary bladder (Renal and urinary disorders) | 3 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 2
Renal impairment (Renal and urinary disorders) | 2 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 3
Malaise (General disorders) | 1 | 1
Oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Cyst (General disorders) | 0 | 1
Face oedema (General disorders) | 1 | 0
Feeling cold (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Thirst (General disorders) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 4 | 5
Gamma-glutamyltransferase increased (Investigations) | 3 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood triglycerides increased (Investigations) | 3 | 0
Blood pressure decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 1
Lipids increased (Investigations) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Rectal polypectomy (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No